CLINICAL TRIAL: NCT00653640
Title: Physical Work Capacity After Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 98-367; R01HD046570 (NIH)
Record Dates: First submitted 2008-04-01; First posted 2008-04-07 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2012-06

CONDITIONS: Traumatic Brain Injury
Keywords: rehabilitation; head injury; 3 months post injury; require manual assistance or walking aids to walk; very slow walking speed; able to follow two step commands
MeSH Terms: conditions — Brain Injuries, Traumatic; Craniocerebral Trauma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): body weight supported treadmill training
  Interventions: Procedure: body weight supported treadmill training
- 2 (Placebo Comparator): traditional physical therapy
  Interventions: Procedure: traditional physical therapy

INTERVENTIONS:
Procedure: body weight supported treadmill training — BWSTT for 12 weeks, 3 times per week
  Arms: 1
Procedure: traditional physical therapy — traditional PT for 12 weeks, 3 times per week
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether body weight supported treadmill training is more effective than traditional physical therapy at restoring gait in persons recovering from traumatic brain injury.

ELIGIBILITY:
Inclusion Criteria:

* traumatic brain injury
* follow two step commands
* between 18 and 60 years old
* between 3 and 36 months post injury

Exclusion Criteria:

* known cardiovascular disease
* uncooperative, behavioral challenges

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2006-05; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Overground gait speed | 12 weeks

SECONDARY OUTCOMES:
aerobic capacity | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kurt A. Mossberg, PT, PhD, Principal Investigator — University of Texas, Galveston
Locations (2):
- United States (2):
  - Transitional Learning Center, Galveston, Texas
  - TIRR Memorial Hermann, Houston, Texas

REFERENCES:
- [Background] Mossberg KA, Ayala D, Baker T, Heard J, Masel B. Aerobic capacity after traumatic brain injury: comparison with a nondisabled cohort. Arch Phys Med Rehabil. 2007 Mar;88(3):315-20. doi: 10.1016/j.apmr.2006.12.006. PMID 17321823
- [Background] Mossberg KA, Greene BP. Reliability of graded exercise testing after traumatic brain injury: submaximal and peak responses. Am J Phys Med Rehabil. 2005 Jul;84(7):492-500. doi: 10.1097/01.phm.0000166883.97562.cd. PMID 15973085
- [Background] Mossberg KA. Reliability of a timed walk test in persons with acquired brain injury. Am J Phys Med Rehabil. 2003 May;82(5):385-90; quiz 391-2. doi: 10.1097/01.PHM.0000052589.96202.BE. PMID 12704280
- [Background] Mossberg KA, Kuna S, Masel B. Ambulatory efficiency in persons with acquired brain injury after a rehabilitation intervention. Brain Inj. 2002 Sep;16(9):789-97. doi: 10.1080/02699050210131894. PMID 12217204
- [Background] Mossberg KA, Masel BE, Gilkison CR, Urban RJ. Aerobic capacity and growth hormone deficiency after traumatic brain injury. J Clin Endocrinol Metab. 2008 Jul;93(7):2581-7. doi: 10.1210/jc.2008-0368. Epub 2008 Apr 15. PMID 18413421
- [Background] Beca SG, High WM Jr, Masel BE, Mossberg KA, Urban RJ. What are critical outcome measures for patients receiving pituitary replacement following brain injury? Pituitary. 2012 Mar;15(1):10-9. doi: 10.1007/s11102-008-0133-3. PMID 18594990
- [Background] Mossberg KA, Amonette WE, Masel BE. Endurance training and cardiorespiratory conditioning after traumatic brain injury. J Head Trauma Rehabil. 2010 May-Jun;25(3):173-83. doi: 10.1097/HTR.0b013e3181dc98ff. PMID 20473091
- [Result] Mossberg KA, Orlander EE, Norcross JL. Cardiorespiratory capacity after weight-supported treadmill training in patients with traumatic brain injury. Phys Ther. 2008 Jan;88(1):77-87. doi: 10.2522/ptj.20070022. Epub 2007 Oct 16. PMID 17940106
- [Result] Mossberg KA, Fortini E. Responsiveness and validity of the six-minute walk test in individuals with traumatic brain injury. Phys Ther. 2012 May;92(5):726-33. doi: 10.2522/ptj.20110157. Epub 2012 Jan 26. PMID 22282772